CLINICAL TRIAL: NCT07238309
Title: A Comparative Study to Evaluate Efficacy of Oversewing Versus Surgical Ligation Clips for Staple Line Reinforcement of the Gastric Pouch to Reduce Post Operative Bleeding in Laparoscopic One Anastomosis Gastric Bypass
Brief Title: Efficacy of Oversewing Versus Surgical Ligation Clips for Staple Line Reinforcement of the Gastric Pouch to Reduce Post Operative Bleeding in Laparoscopic One Anastomosis Gastric Bypass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Gamal Abd Elghany, General and Laparoscopic surgeon, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: laparoscopic gastric bypass
Record Dates: First submitted 2025-09-18; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Gastric Bypass Surgery
Keywords: Laparoscopic One Anastomosis Gastric Bypass surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Through-and-through sutures (Experimental): through-and-through sutures with 3-0 absorbable monofilament sutures will be used .
  Interventions: Procedure: Oversewing
- Titanium Ligation clips (Experimental): Titanium Ligation clips will be used .
  Interventions: Procedure: Surgical Ligation Clips

INTERVENTIONS:
Procedure: Oversewing — Through-and-through sutures with 3-0 absorbable monofilament sutures will be placed over the staple line to reinforce it in laparoscopic one anastomosis gastric bypass surgery.
  Arms: Through-and-through sutures
Procedure: Surgical Ligation Clips — Titanium Ligation clips will be used to secure hemostasis and reinforce staple line by approximating tissue edges in laparoscopic one anastomosis gastric bypass surgery.
  Arms: Titanium Ligation clips

SUMMARY:
1. To test if there is a significant differences between Oversewing versus surgical ligation clips for staple line reinforcement of the gastric pouch regarding the reduction of post operative bleeding and the need for blood transfusions in laparoscopic one anastomosis gastric bypass.
2. To assess whether oversewing or the use of surgical clips is more effective in reducing operative time and Cost analysis in (OAGB).
3. To Provide evidence-based recommendations on staple line reinforcement techniques in OAGB, emphasizing patient safety and procedural efficiency

DETAILED DESCRIPTION:
Obesity is a disease related to reduced life expectancy, as well as increased morbidity and mortality. In recent years, bariatric surgery has become an increasingly widespread form of treatment for severe obesity and its associated diseases . The increased spread of bariatric surgery is associated with its long-term reliability and also its high cost-benefit ratio.

According to the International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO) registry (calendar years 2014-2018), there are three main surgical procedures in common use: sleeve gastrectomy (SG), Roux-en-Y gastric bypass (RYGB) and laparoscopic one anastomosis gastric bypass (OAGB) . OAGB, introduced by Rutledge in 1997 is a restrictive and malabsorptive bariatric surgical procedure and is the fourth most performed bariatric technique in Europe and in the Asia/Pacific area, with an increasing trend .

In the last 15 years, several authors have demonstrated the effectiveness of this surgical technique in terms of both weight loss and the resolution of comorbidities, especially type 2 diabetes mellitus (T2DM).

Despite the described advantages, LSG still conveys some risks. Early staple line complications, such as bleeding and leaks, may occur, and their incidence may vary from 1 to 6% . Such complications can be devastating and life-threatening. Besides, they entail additional healthcare-related costs. It has been proposed that staple line complications can be reduced by staple line reinforcement (SLR).

Staple line reinforcement (SLR) has been proposed to decrease the risk of these complications by several options: oversewing the staple line with a running absorbable suture, buttressing it with specific materials or roofing the staple line. Although it has been postulated that there are fewer complications, SLR remains controversial and its effectiveness is still unclear . Some surgeons still have concerns about SLR, either because of Uncertainty about its benefits and/or its financial costs. Moreover, it has been argued that oversewing itself could carry additional risks. The potential for leakage and bleeding could increase due to tearing at the suture penetration point, and the running suture may lead to sleeve stricture and tissue ischemia.

Two common techniques for this purpose are oversewing and the use of surgical ligation clips. Oversewing involves suturing over the staple line, which has been shown to significantly reduce the incidence of staple line bleeding, with rates dropping from 9-13.7% to as low as 1.4-2%, While effective and cost-efficient.

Oversewing can increase operative time due to the additional suturing required .

On the other hand, surgical ligation clips provide a rapid method for achieving hemostasis and reinforcing the staple line. Research indicates that ligation clips are effective in controlling bleeding, with low complication rates (e.g., only 1.7% episodes of melena reported).

Both techniques demonstrate comparable efficacy in preventing complications, and the choice between them may depend on clinical context, surgeon preference, and resource availability. Further studies comparing long-term outcomes would enhance understanding of their relative effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* ✔ Age ≥ 18years old

  * Sex: both sex
  * Fit for bariatric surgery
  * body mass index (BMI) of 40 kg/m 2 or higher or BMI between 35 and 40 kg/m2 with significant comorbidities, such as T2DM, hypertension, OSAS or significant osteo- articular alterations, not responsive to medical therapies
  * Patients should have tried and failed to lose weight using diet, exercise, and/or medication for at least 6 months
  * Patients or first guardians accept to participate in the current study
  * Patients or first guardians accept to provide informed written consent

Exclusion Criteria:

* Patients less than 18 years old

  * Patients or first guardians refused to participate in the current study
  * Patients or first guardians refused to provide informed written consent
  * All patients with bleeding disorders and patients needing re-exploration for bleeding other than staple line Pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Clinically Significant Postoperative Bleeding Within 30 Days | 30 days after laparoscopic one-anastomosis gastric bypass surgery
  Proportion of participants experiencing clinically significant postoperative bleeding within 30 days of laparoscopic one-anastomosis gastric bypass.
  Clinically significant postoperative bleeding is defined as the occurrence of any of the following events within 30 days after surgery:
  1. Re-operation for bleeding,
  2. Endoscopic or radiologic intervention to control bleeding,
  3. Transfusion of ≥ 1 unit of packed red blood cells for acute postoperative blood loss, or
  4. Hemoglobin drop ≥ 2.0 g/dL from immediate postoperative baseline accompanied by hemodynamic instability (systolic blood pressure < 90 mmHg or requiring vasopressor support).
  The analysis metric will be the number and percentage of participants (n, %) with at least one bleeding event in each treatment arm. Between-group comparison will use the risk difference with 95 % confidence interval (or the pre-specified statistical test per the statistical analysis plan).

SECONDARY OUTCOMES:
Operative Time | Intraoperative (recorded during procedure)
  Duration of surgery measured in minutes from skin incision to skin closure. Analysis metric: mean (SD) operative time per group; compared using pre-specified statistical tests.

CONTACTS AND LOCATIONS:
Overall Officials: George AbdElFady Nashed Aiad, M.D, Principal Investigator — professor in General and Laparoscopic surgery
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Background] Wolfe BM, Kvach E, Eckel RH. Treatment of Obesity: Weight Loss and Bariatric Surgery. Circ Res. 2016 May 27;118(11):1844-55. doi: 10.1161/CIRCRESAHA.116.307591. PMID 27230645